CLINICAL TRIAL: NCT05685537
Title: Impact of Levosimendan Preconditioning on Critical Care and In-hospital Lengths of Stay After Cardiac Surgery With Bypass Surgery
Acronym: LevoCCV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Klein Thomas, Medical Doctor, Central Hospital, Nancy, France
Other Study IDs: 2022_PI_118
Record Dates: First submitted 2022-12-20; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-12

CONDITIONS: Levosimendan; Cardiac Surgery; Cardiopulmonary Bypass
MeSH Terms: interventions — Simendan; Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Levosimendan - Interventional: Major patients in heart failure with impaired LVEF (< 40%) who have undergone left heart surgery (coronary artery bypass grafting and/or mitral and/or aortic valve replacement) under extracorporeal circulation between 01/01/2018 and 28/02/2022 at the Nancy University Hospital or at the University Hospital of Rennes, Rouen or Amiens, and who have received Levosimendan preoperatively
  Interventions: Drug: Levosimendan
- Non Levosimendan - Control: Major patients in heart failure with impaired LVEF (< 40%) who have undergone left heart surgery (coronary artery bypass grafting and/or mitral and/or aortic valve replacement) under extracorporeal circulation between 01/01/2018 and 28/02/2022 at the Nancy University Hospital or at the University Hospital of Rennes, Rouen or Amiens, and who have not received Levosimendan preoperatively

INTERVENTIONS:
Drug: Levosimendan — Initiation of levosimendan 48 hours before surgery
  Other Names: Interventional
  Groups: Levosimendan - Interventional

SUMMARY:
Levosimendan, a drug with inotropic, vasodilatory and myocardial protective properties, has been proposed for the prevention and treatment of postoperative low cardiac output syndrome in cardiac surgery. Despite preliminary studies with promising results, large randomized controlled trials aimed at demonstrating the benefits of levosimendan did not show superiority over placebo in this indication. However, in these studies, the infusion was neither performed at the maximum dosage nor during the 24 hours preceding the surgery, but mainly at the very beginning of the operation. However, post hoc analyses showed a reduction in mortality and in the occurrence of low cardiac output syndrome in the subgroup of patients who had undergone isolated coronary artery bypass grafting, in contrast to those who had undergone valvular or combined surgery. Another recent study suggests that under similar conditions, preconditioning with levosimendan started 48 hours before surgery reduces the length of stay in intensive care and the average cost of hospitalization. There are no formal recommendations on the prophylactic use of levosimendan in cardiac surgery for heart failure patients with impaired LVAS. However, the France-Levo registry, a multicenter observational study requested by the HAS, has shown that in real practice there is a place for preconditioning with levosimendan, which is used in this indication for 7% of the patients in the registry. The Cardiovascular Surgery and Transplantation Department of the Nancy Brabois University Hospital, which actively participated in the France-Levo registry, is one of the cardiac surgery centers that uses this practice, as is the University Hospital of Rouen. It is interesting to be able to evaluate retrospectively whether levosimendan preconditioning has a positive impact on the postoperative prognosis of patients and more particularly on the reduction of the length of stay in critical care and in hospital compared to standard management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure impaired LVEF (< 40%), who have undergone left heart surgery (coronary artery bypass grafting and/or mitral and/or aortic valve replacement) under extracorporeal circulation between 01/01/2018 and 28/02/2022 at the Nancy University Hospital or the University Hospital of Rennes, Rouen or Amiens

Exclusion Criteria:

* Initiation of levosimendan > 48 hours or < 24 hours before surgery
* ECMO pre- or post-op

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Preoperative heart failure patients with impaired LVEF who underwent left heart surgery (coronary artery bypass grafting and/or mitral and/or aortic valve replacement) under extracorporeal circulation from 01/09/2018 to 28/02/2022 at the CHRU de Nancy, CHRU de Rennes, CHRU de Rouen or CHRU d'Amiens.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Length of stay in ICU | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 3 months
  To evaluate the impact of levosimendan preconditioning preoperatively for cardiac surgery on critical care length of stay in patients with heart failure with impaired preoperative LVAS.

SECONDARY OUTCOMES:
On 1-year mortality | 1 year after Levosimendan exposure
  To evaluate the impact of preconditioning with Levosimendan before cardiac surgery in patients with heart failure and impaired left ventricular dysfunction on 1-year mortality
the total length of hospital stay | start date of hospitalization in intensive care to the date of discharge from conventional sectors evaluated up to 3 months
  To evaluate the impact of preconditioning with Levosimendan preoperatively for cardiac surgery in patients with heart failure with impaired preoperative left ventricular dysfunction on the total length of hospital stay
left ventricular systolic function at hospital discharge | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 3 months
  To evaluate the impact of Levosimendan preconditioning before cardiac surgery in patients with heart failure and impaired on left ventricular systolic function at hospital discharge
duration of catecholamine use after surgery | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 3 months
  To evaluate the impact of preconditioning with Levosimendan before cardiac surgery in patients with heart failure and impaired left ventricular function before surgery on the duration of catecholamine use after surgery
severity of postcardiotomy cardiogenic shock and/or postoperative vasoplegia using the score Vasoactive Inotropic Score (VIS) | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 3 months
  To evaluate the impact of preconditioning with Levosimendan in preoperative cardiac surgery in patients with heart failure with impaired preoperative LVAS on the severity of postcardiotomy cardiogenic shock and/or postoperative vasoplegia
acute renal failure postoperatively | on discharge from the intensive care unit
  To evaluate the impact of preconditioning with Levosimendan preoperatively for cardiac surgery in patients with heart failure with impaired left ventricular function preoperatively on the rate of acute renal failure postoperatively
readmission rate for cardiac decompensation | within one year of Levosimendan administration
  To evaluate the impact of preconditioning with Levosimendan preoperatively for cardiac surgery in patients with heart failure and impaired LVAS preoperatively on the readmission rate for cardiac decompensation

CONTACTS AND LOCATIONS:
Overall Officials: KLEIN Thomas, MD, Principal Investigator — Intensive care unit
Locations (1):
- 'CHRU Nancy, Vandœuvre-lès-Nancy, Meurthe Et Moselle, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erb J, Beutlhauser T, Feldheiser A, Schuster B, Treskatsch S, Grubitzsch H, Spies C. Influence of levosimendan on organ dysfunction in patients with severely reduced left ventricular function undergoing cardiac surgery. J Int Med Res. 2014 Jun;42(3):750-64. doi: 10.1177/0300060513516293. Epub 2014 Apr 29. PMID 24781725
- [Background] Sanfilippo F, Knight JB, Scolletta S, Santonocito C, Pastore F, Lorini FL, Tritapepe L, Morelli A, Arcadipane A. Levosimendan for patients with severely reduced left ventricular systolic function and/or low cardiac output syndrome undergoing cardiac surgery: a systematic review and meta-analysis. Crit Care. 2017 Oct 19;21(1):252. doi: 10.1186/s13054-017-1849-0. PMID 29047417
- [Background] van Diepen S, Mehta RH, Leimberger JD, Goodman SG, Fremes S, Jankowich R, Heringlake M, Anstrom KJ, Levy JH, Luber J, Nagpal AD, Duncan AE, Argenziano M, Toller W, Teoh K, Knight JD, Lopes RD, Cowper PA, Mark DB, Alexander JH. Levosimendan in patients with reduced left ventricular function undergoing isolated coronary or valve surgery. J Thorac Cardiovasc Surg. 2020 Jun;159(6):2302-2309.e6. doi: 10.1016/j.jtcvs.2019.06.020. Epub 2019 Jun 21. PMID 31358329
- [Background] Cholley B, Caruba T, Grosjean S, Amour J, Ouattara A, Villacorta J, Miguet B, Guinet P, Levy F, Squara P, Ait Hamou N, Carillion A, Boyer J, Boughenou MF, Rosier S, Robin E, Radutoiu M, Durand M, Guidon C, Desebbe O, Charles-Nelson A, Menasche P, Rozec B, Girard C, Fellahi JL, Pirracchio R, Chatellier G; -. Effect of Levosimendan on Low Cardiac Output Syndrome in Patients With Low Ejection Fraction Undergoing Coronary Artery Bypass Grafting With Cardiopulmonary Bypass: The LICORN Randomized Clinical Trial. JAMA. 2017 Aug 8;318(6):548-556. doi: 10.1001/jama.2017.9973. PMID 28787507
- [Result] Levin R, Degrange M, Del Mazo C, Tanus E, Porcile R. Preoperative levosimendan decreases mortality and the development of low cardiac output in high-risk patients with severe left ventricular dysfunction undergoing coronary artery bypass grafting with cardiopulmonary bypass. Exp Clin Cardiol. 2012 Sep;17(3):125-30. PMID 23620700